CLINICAL TRIAL: NCT05885672
Title: A Multi-Modal Approach to Improving the Early Detection of Cardiometabolic Disease Risk
Brief Title: Improving the Early Detection of Cardiometabolic Disease Risk
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern Mississippi (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0446
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Capillary and intravenous blood collection for the analysis of:
  * Glucose
  * Insulin
  * Blood Lipids
  * Inflammatory biomarkers (tumor necrosis factor-a)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Adults: Adults between the ages of 18 and 39 years
  Interventions: Behavioral: Online psychoeducational lifestyle intervention

INTERVENTIONS:
Behavioral: Online psychoeducational lifestyle intervention — A webpage-baed intervention focused on lifestyle interventions that aim to reduce metabolic syndrome severity.

SUMMARY:
The goal of this observational study is to reduce an individual's cardiometabolic disease risk by improving the ability to detect cardiometabolic disease risk in young adults through the use of novel technologies that increase access to and examine the utility of, a continuous metabolic syndrome severity score. An additional goal of this study is to understand the barriers to engagement in health-promoting behaviors and beliefs about interventions aimed at mitigating metabolic syndrome risk through a brief online lifestyle intervention.

The main question[s] it aims to answer are:

* Can a smartphone-based imaging system accurately predict a continuous metabolic syndrome severity score, in addition to other markers of cardiometabolic disease, in young adults?
* What is the relationship between autonomic dysfunction and metabolic syndrome severity in a cohort of young adults?
* What is the relationship between peripheral vascular dysfunction and metabolic syndrome severity in a cohort of young adults?
* What are the associations between metabolic syndrome severity and gait and functional ability in young adults using novel markerless motion capture technology?
* What are the attitudes and barriers towards lifestyle interventions targeted to reduce metabolic syndrome severity?
* What are the treatment-seeking and willingness to engage behaviors toward a webpage focused on lifestyle interventions to reduce metabolic syndrome severity?

Participants will be asked to undergo several assessments across four separate days which are design designed to determine the associations between cardiometabolic health markers and components of:

* body composition
* cardiovascular function
* functional ability
* attitudes and behaviors towards health-related interventions

ELIGIBILITY:
Inclusion Criteria:

- adults between the ages of 18-39 years of age

Exclusion Criteria:

* Younger than 18 or older than 39
* Pregnant
* Breastfeeding or lactating
* Missing any limbs or part of a limb
* Having a substantial amount of metal implants (metal plates or complete joint replacements)
* Having a pacemaker or any other electrical implant
* Type I diabetes
* Gestational diabetes
* Taking insulin
* Diagnosed heart failure, cardiomyopathy (dilated or hypertrophic), valvular disease
* Any history of severe traumatic brain injury or mild traumatic brain injury within the last two years
* Kidney disease
* Liver disease
* Thyroid disease
* Any diagnosed neurological or neurodegenerative diseases
* Having received ionizing radiation from a medical procedure within the last 30 days
* Being on a medically prescribed diet
* Having donated blood or plasma in the last 20 days prior to blood collection procedures
* Taking any supplements/medications that may interfere with the results of the study
* Any injury or physical impairment that would prevent performing any functional measures for this study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults between the ages of 18 and 39 with or without metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline
  Resting systolic and diastolic blood pressure
Waist Circumference | Baseline
  Circumference of the waist measured by tape measure at the level of the iliac crest
Fasting blood glucose | Baseline
  Blood glucose collected from capillary blood
Blood lipids | Baseline
  Triglycerides, total cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol collected from capillary blood
Metabolic syndrome severity score | Baseline
  A race and sex-specific equation that uses systolic blood pressure, waist circumference, and blood lipids to calculate a single continuous score that quantifies a person's overall cardiometabolic disease severity on a continuum where higher scores equal a worse outcome and negative scores equal a better outcome. The scale does not have bound and is infinite in positive and negative directions.
Insulin | Baseline
  Insulin collected from intravenous blood
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Baseline
  Equation that estimates insulin resistance from glucose and insulin measurements
Tumor necrosis factor-alpha | Baseline
  Common biomarker of systemic inflammation collected from intravenous blood
Body fat percentage | Baseline
  The percentage of body fat estimated using smartphone-based digital imaging and near-infrared reactance spectroscopy
Fat mass | Baseline
  The weight of fat mass in kilograms estimated using smartphone-based digital imaging and near-infrared reactance spectroscopy
Fat-free mass | Baseline
  The weight of fat-free mass in kilograms estimated using smartphone-based digital imaging and near-infrared reactance spectroscopy
Body circumferences | Baseline
  Central (trunk) and segmental (arms and legs) circumference estimated using smartphone-based digital imaging
Heart Rate Variability | Baseline
  Index of cardiac autonomic control collected via one-lead electrocardiogram
Cardiac Baroreflex Sensitivity | Baseline
  Measure of parasympathetic and sympathetic regulation collected via one-lead electrocardiogram and finger photoplethysmography
Flow-mediated changes in vascular diameter | Baseline
  Changes in vascular diameter during 5 minutes of post-occlusive reactive hyperemia collected via duplex Doppler ultrasound
Flow-mediated changes in blood flow | Baseline
  Changes in blood flow during 5 minutes of post-occlusive reactive hyperemia collected via duplex Doppler ultrasound
Flow-mediated changes in blood pressure | Baseline
  Changes in blood pressure during 5 minutes of post-occlusive reactive hyperemia collected via finger photoplethysmography
Flow-mediated changes in vascular conductance | Baseline
  Changes in vascular conductance during 5 minutes of post-occlusive reactive hyperemia calculated as flow per unit of blood pressure
Flow-mediated changes in vascular resistance | Baseline
  Changes in vascular resistance during 5 minutes of post-occlusive reactive hyperemia calculated as blood pressure per unit of flow
Flow-mediated changes in skeletal muscle oxygenation | Baseline
  Changes in skeletal muscle oxygenated/deoxygenated hemoglobin saturation during 5 minutes of post-occlusive reactive hyperemia collected via near-infrared spectroscopy
Passive Limb Movement Mediated Changes in Vascular Diameter | Baseline
  Changes in vascular diameter during passive limb movement collected via duplex Doppler ultrasound
Passive Limb Movement Mediated Changes in Blood Flow | Baseline
  Changes in blood flow during passive limb movement collected via duplex Doppler ultrasound
Passive Limb Movement Mediated Changes in Blood Pressure | Baseline
  Changes in blood pressure during passive limb movement collected via finger photoplethysmography
Passive Limb Movement Mediated Changes in Vascular Conductance | Baseline
  Changes in vascular conductance during passive limb movement calculated as flow per unit of pressure
Passive Limb Movement Mediated Changes in Vascular Resistance | Baseline
  Changes in vascular resistance during passive limb movement calculated as the pressure per unit of flow
Passive Limb Movement Mediated Changes in Skeletal Muscle Oxygenation | Baseline
  Changes in skeletal muscle oxygenation during passive limb movement collected via near-infrared spectroscopy
Carotid-Femoral Pulse Wave Velocity | Baseline
  Index of arterial stiffness collected during rest collected via applanation tonometry and auscultation based wave analysis
Cold Pressor Test Blood Pressure Responses | Baseline
  Changes in blood pressure during three minutes of cold-pressor activation collected via finger photoplethysmography
Cold Pressor Test Heart Rate Responses | Baseline
  Changes in heart rate during three minutes of cold-pressor activation collected via one-lead electrocardiogram
Cold Pressor Test Vascular Conductance Responses | Baseline
  Changes in vascular conductance during three minutes of cold-pressor activation calculated as flow per unit of pressure
Cold Pressor Test Vascular Resistance Responses | Baseline
  Changes in vascular resistance during three minutes of cold-pressor activation calculated as pressure per unit of flow
Cold Pressor Test stroke volume Responses | Baseline
  Changes in stroke volume during three minutes of cold-pressor activation collected via finger photoplethysmography or duplex Doppler ultrasound
Cold Pressor Test Cardiac Output Responses | Baseline
  Changes in cardiac output during three minutes of cold-pressor activation collected via finger photoplethysmography or duplex Doppler ultrasound
Metaboreflex Blood Pressure Responses | Baseline
  Changes in blood pressure during rhythmic handgrip exercise with graded blood flow restriction (minutes 0, 2, 4, 6, and 8) collected via finger photoplethysmography
Metaboreflex Heart Rate Responses | Baseline
  Changes in heart rate during rhythmic handgrip exercise with graded blood flow restriction (minutes 0, 2, 4, 6, and 8) collected via one-lead electrocardiogram
Metaboreflex Vascular Conductance Responses | Baseline
  Changes in vascular conductance during rhythmic handgrip exercise with graded blood flow restriction (minutes 0, 2, 4, 6, and 8) calculated as flow per unit of pressure
Metaboreflex Vascular Resistance Responses | Baseline
  Changes in vascular resistance during rhythmic handgrip exercise with graded blood flow restriction (minutes 0, 2, 4, 6, and 8) calculated as pressure per unit of flow
Metaboreflex Stroke Volume Responses | Baseline
  Changes in stroke volume during rhythmic handgrip exercise with graded blood flow restriction (minutes 0, 2, 4, 6, and 8) collected via finger photoplethysmography or duplex Doppler ultrasound
Metaboreflex Cardiac Output Responses | Baseline
  Changes in cardiac output during rhythmic handgrip exercise with graded blood flow restriction (minutes 0, 2, 4, 6, and 8) collected via finger photoplethysmography or duplex Doppler ultrasound
Functional Sympatholysis Blood Flow Responses | Baseline
  Changes in limb blood flow during three minutes of cold-pressor activation with superimposed rhythmic handgrip exercise Collected via finger photoplethysmography
Functional Sympatholysis Vascular Conductance Responses | Baseline
  Changes in vascular conductance during three minutes of cold-pressor activation with superimposed rhythmic handgrip exercise calculated as flow per unit of pressure
Functional Sympatholysis Vascular Resistance Responses | Baseline
  Changes in vascular resistance during three minutes of cold-pressor activation with superimposed rhythmic handgrip exercise Calculated as pressure per unit of flow
Functional Sympatholysis Blood Pressure Responses | Baseline
  Changes in blood pressure during three minutes of cold-pressor activation with superimposed rhythmic handgrip exercise collected via finger photoplethysmography
Gait velocity | Baseline
  Self-selected walking velocity over level ground measured with a timing gate system.
Gait velocity | Immediately post 6-minute walk test
  Self-selected walking velocity over level ground measured with a timing gate system.
Stride Length | Baseline
  Length of stride, measured as the lateral distance between feet during walking measured with a motion capture system.
Stride Length | Immediately post 6-minute walk test
  Length of stride, measured as the lateral distance between feet during walking measured with a motion capture system.
Stride Width | Baseline
  Width of stride, measured as the lateral distance between feet during walking measured with a motion capture system.
Stride Width | Immediately post 6-minute walk test
  Width of stride, measured as the lateral distance between feet during walking measured with a motion capture system.
Gait Cadence | Baseline
  Steps taken per minute measured with a motion capture system.
Gait Cadence | Immediately post 6-minute walk test
  Steps taken per minute measured with a motion capture system.
Ankle joint angle | Baseline
  Ankle angle during level ground walking measured in degrees measured with a motion capture system.
Ankle joint moment | Baseline
  Ankle moment during level ground walking measured in newton-meters measured with a motion capture system.
Ankle joint angle | Immediately post 6-minute walk test
  Ankle angle during level ground walking measured in degrees measured with a motion capture system.
Ankle joint moment | Immediately post 6-minute walk test
  Ankle moment during level ground walking measured in newton-meters measured with a motion capture system.
Knee joint angle | Baseline
  Knee angle during level ground walking measured in degrees measured with a motion capture system.
Knee joint moment | Baseline
  Knee moment during level ground walking measured in newton-meters measured with a motion capture system.
Knee joint angle | Immediately post 6-minute walk test
  Knee angle during level ground walking measured in degrees measured with a motion capture system.
Knee joint moment | Immediately post 6-minute walk test
  Knee moment during level ground walking measured in newton-meters measured with a motion capture system.
Hip joint angle | Baseline
  Hip angle during level ground walking measured in degrees measured with a motion capture system.
Hip joint moment | Baseline
  Hip moment during level ground walking measured in newton-meters measured with a motion capture system.
Hip joint angle | Immediately post 6-minute walk test
  Hip angle during level ground walking measured in degrees measured with a motion capture system.
Hip joint moment | Immediately post 6-minute walk test
  Hip moment during level ground walking measured in newton-meters measured with a motion capture system.
Ground reaction forces | Baseline
  Three-dimensional ground reaction forces during level ground walking measured with a motion capture system.
Ground reaction forces | Immediately post 6-minute walk test
  Three-dimensional ground reaction forces during level ground walking measured with a motion capture system.
Center of pressure - right leg | Baseline
  Whole body center of pressure displacement
Center of pressure - left leg | Baseline
  Whole body center of pressure displacement
Center of pressure - bilateral | Baseline
  Whole body center of pressure displacement
Timed-up and go | Baseline
  Time (seconds) for participant to stand up from chair, walk 3 meters, and return
Sit-to-stand | Baseline
  Time (seconds) for participant to stand up from chair and sit back down (5 repetitions)
Time Up and Down Stairs | Baseline
  Time (seconds) for participant to stand ascend and descend a single flight (10 steps) of stairs
Isometric strength | Baseline
  Isometric muscle strength of hip flexors and extensors, knee flexors and extensors, and ankle dorsi- and plantar flexors of the right leg
Visceral adipose tissue | Baseline
  Absolute fat-mass around the visceral organs in kilograms measured using dual-energy x-ray absorptiometry and near-infrared reactance spectroscopy
Subcutaneous adipose tissue | Baseline
  Absolute fat-mass under the cutaneous layer of the skin in kilograms measured using dual-energy x-ray absorptiometry
Motivation and Attitudes Towards Health | Baseline
  Motivation and Attitudes Towards Changing Health Scale. Scores range from 5-45, which higher scores indicating higher motivation and more positive attitudes towards changing health behavior
Readiness for Behavior Change | Baseline
  Readiness for Change Questionnaire. Separate subscales are calculated for each of the 5 stages of change (pre-contemplation, contemplation, preparation, action, maintenance) with higher scores indicating a greater likelihood of an individual being in that stage of change versus another. The 12 items on this scale are scored on a scale of -2 to +2 (-2 = Strongly disagree, -1 Disagree, 0 = Unsure, +1 = Agree, +2 = Strongly Agree).
Treatment Seeking Behavior | Baseline
  Whether participant engages with educational webpage about health behavior change. This is a dichotomous yes/no value based on whether someone clicks on the webpage or not.

SECONDARY OUTCOMES:
Height | Baseline
  Height collected using a stadiometer
Weight | Baseline
  Weight collected using a stadiometer

CONTACTS AND LOCATIONS:
Overall Officials: Austin J Graybeal, PhD, Principal Investigator — University of Southern Mississippi; Jon Stavres, PhD, Principal Investigator — University of Southern Mississippi; Tanner Thorsen, PhD, Principal Investigator — University of Southern Mississippi; Megan Renna, PhD, Principal Investigator — University of Southern Mississippi
Locations (1):
- University of Southern Mississippi - School of Kinesiology and Nutrition, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data and analytic code to be made available using Open Science Framework
Supporting Information: SAP, Analytic Code
Time Frame: Upon publication of the primary results and will be kept available for 18 months

REFERENCES:
- [Derived] Graybeal AJ, Compton AT, Swafford SH, Brandner CF, Thorsen T, Renna ME, Stavres J. Measurements of Abdominal Obesity are Associated with Metabolic Syndrome Severity Independent of Hypertensive Phenotype in White but not Black Young Adults. J Racial Ethn Health Disparities. 2025 Aug;12(4):2299-2311. doi: 10.1007/s40615-024-02051-8. Epub 2024 Jun 20. PMID 38902464